CLINICAL TRIAL: NCT03993769
Title: CSD190101: An Unblinded, Randomized, Multi-site, Two-way Crossover Study to Assess Nicotine Pharmacokinetic Parameters After Use of Two Smokeless Tobacco Products A19010-F and B19010-F in Healthy Adult Snus Consumers.
Brief Title: CSD190101: A Study to Assess Nicotine Pharmacokinetic Parameters After Use of Two Smokeless Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD190101
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A19010-F, B19010-F Use Group (Experimental): Use of product A19010-F exclusively for 4 days prior to a PK assessment for plasma nicotine concentrations, followed by use of product B19010-F exclusively for 4 days prior to a PK assessment for plasma nicotine concentrations.
  Interventions: Other: A19010-F; Other: B19010-F
- B19010-F, A19010-F Use Group (Experimental): Use of product B19010-F exclusively for 4 days prior to a PK assessment for plasma nicotine concentrations, followed by use of product A19010-F exclusively for 4 days prior to a PK assessment for plasma nicotine concentrations.
  Interventions: Other: A19010-F; Other: B19010-F

INTERVENTIONS:
Other: A19010-F — A snus product
Other: B19010-F — A snus product

SUMMARY:
The purpose of this study is to compare plasma nicotine uptake in adult snus consumers after using investigational snus products (A19010-F and B19010-F).

DETAILED DESCRIPTION:
This will be an unblinded, randomized, multi-site, two-way crossover study to assess nicotine pharmacokinetic parameters after use of two smokeless tobacco products A19010-F and B19010-F in healthy adult snus consumers. Eligible subjects will be confined to the site for 9 days and randomized to one of two investigational product (IP) (A: A19010-F and B: B19010-F) use sequences (AB/BA). Each subject will use a single product exclusively for 4 days prior to a PK assessment for plasma nicotine concentrations, and then subjects will use the other product exclusively for 4 days prior to a PK assessment for plasma nicotine concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires;
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of signing the ICF;
3. Positive urine cotinine test at the Screening Visit and Day 1;
4. Childbearing females must be willing to use a form of contraception acceptable to the Principal Investigator (PI) from the time of signing the ICF until study discharge; acceptable methods include:

   a. Female subjects who are heterosexually active and of childbearing potential (e.g., neither surgically sterile postmenopausal) must have been using one of the following forms of contraception for the time period indicated and agree to continue using it through completion of the study:
   * Hormonal (e.g., oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to Check-in
   * Double barrier (i.e., condom with spermicide or diaphragm with spermicide) consistently for at least 4 weeks prior to Check-in
   * Intrauterine device for at least 4 months prior to Check-in
   * Exclusive partner who has been vasectomized for at least 6 months (inclusive) prior to Check-in
   * Female subjects of childbearing potential who are not currently engaging
   * In heterosexual intercourse must agree to use one of the above methods of birth control through completion of study, in the event that they have heterosexual intercourse during the course of the study.
5. Female subjects who are of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Check in:

   * Hysteroscopic sterilization (including Essure® or similar nonsurgical sterilization procedures);
   * Bilateral tubal ligation or bilateral salpingectomy
   * Hysterectomy
   * Bilateral oophorectomy
6. Subjects' primary tobacco product must be a mint or mint-like flavor of snus. Poly use of other (non-snus) forms of tobacco- and/or nicotine-containing products will be allowed if frequency of use of other products is less than or equal to four days per week (e.g., vaping) OR less than or equal to 15 cigarettes per week.
7. Self-reports currently using at least one container of their usual brand (UB) snus per week for at least 3 months prior to randomization;
8. Agrees to exclusively use the IP and not use any other tobacco- or nicotine-containing product during the study;
9. Willing to comply with the requirements of the study;
10. Able to safely perform the required study procedures, as determined by the PI.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, chronic pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study;
2. History, presence of, or clinical laboratory test results indicating diabetes;
3. Hemoglobin level < 11.0 g/dL for females and < 12.0 g/dL for males at the Screening Visit;
4. History or presence of bleeding or clotting disorders;
5. Daily use of aspirin (> 325mg/day) or anticoagulants;
6. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing the ICF;
7. Plasma donation within (≤) 7 days of signing the ICF;
8. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for 5 minutes;
9. Weight of ≤ 110 pounds;
10. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV);
11. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that have been surgically and/or cryogenically removed;
12. Use of any medication or substance that aids in smoking cessation, including but not limited to any NRT (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to signing the ICF;
13. Participation in another clinical trial within (≤) 30 days of signing the ICF (the 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study);
14. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the study;
15. A positive urine drug screen without evidence of prescribed corresponding acceptable concomitant medication(s) at the Screening Visit or at check-in on Day 1;
16. Postponing a decision to quit using tobacco- or nicotine-containing products to participate in this study or a previous quit attempt within (≤) 30 days prior to signing the ICF;
17. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol breathalyzer result at the Screening Visit and check-in on Day 1;
18. Employed by a tobacco- or other nicotine-product manufacturing company, or the study site, or handles tobacco- or nicotine-containing products as part of their job;
19. Presence of gum bleeding and/or abscess, open mouth sores or oral ulcers at Screening, Check-in, or prior to Day 5 product use (just prior to switching IP);
20. Full dentures or braces (with the exception of night guard/retainer, and dental implants which may be allowed; if subjects is missing all lower teeth and does not use dentures will also be allowed);
21. Determined by the PI to be inappropriate for the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
AUCnic 0-240 | 240 minutes
  Area under the baseline-adjusted nicotine concentration-versus-time curve from time zero to 240 minutes after the start of a 30-minute single IP use period.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hong, MD, Study Director — RAIS
Locations (6):
- United States (6):
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - Central Kentucky Research, Lexington, Kentucky
  - QPS Bio-Kinetic, Springfield, Missouri
  - High Point Clinical Trials Center, High Point, North Carolina
  - New Orleans Center for Clinical Research (NOCCR), Knoxville, Tennessee
  - Spaulding Clinical Research, LLC, West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: No